CLINICAL TRIAL: NCT06438510
Title: A Pilot Study to Evaluate the Impact of Gastric Mucosal Ablation (GMA) of the Fundus With Hybrid Argon Plasma Coagulation (HybridAPC) Combined With Endoscopic Sleeve Gastroplasty (ESG) on Obesity
Brief Title: The Fulness Trial (Fundus mUcosaL abLation aNd Endoscopic Sleeve Gastroplasty)
Acronym: FULNESS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, BOSKOSKI IVO, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5646
Record Dates: First submitted 2023-06-15; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm (Experimental): All patients undergo Endoscopic Sleeve Gastroplasty (ESG) and HybridAPC. ESG will be performed using a flexible endoscopic suturing system (OverStitchTM; Apollo Endosurgery, Austin, TX, USA) connected to a gastroscope. Full- thickness sutures will be placed from the angulus to the gastric fundus using a U-shaped pattern with 2.0 nonabsorbable suture thread. Biopsy tissue will be collected from the gastric fundus and the samples will be fixed for histopathologic examination. HybridAPC is an highly controlled mucosal lift applied by the waterjet function and the subsequent thermal ablation applied by APC. First the fluid cushion is injected into submucosa until a size in the range of 2 - 3 cm is achieved (pressure setting of E20 up to E 30). Second the mucosa is being ablated on the surface of this fluid cushion (30 - 50 Watts, argon gas flow 0.8 L/min)
  Interventions: Procedure: Gastric Mucosal Ablation (GMA) of the fundus with Hybrid Argon Plasma Coagulation (HybridAPC) combined with Endoscopic Sleeve Gastroplasty (ESG)

INTERVENTIONS:
Procedure: Gastric Mucosal Ablation (GMA) of the fundus with Hybrid Argon Plasma Coagulation (HybridAPC) combined with Endoscopic Sleeve Gastroplasty (ESG) — All endoscopic procedures will be performed with the patient in the supine position, under general anesthesia, with endotracheal intubation, in CO2 using a flexible endoscopic suturing system (OverStitchTM; Apollo Endosurgery, Austin, TX, USA) connected to a dual-channel endoscope (GIF-2TH180 or GIF-2TH160; Olympus, Center Valley, PA, USA ). The HybridAPC with submucosal injection and APC will be delivered by ErbeJet®2. ESG will be obtained by placing full-thickness sutures in the body gastric wall, from the angulus to the gastric fundus. Biopsy tissue will be collected from the gastric fundus and the samples will be fixed for histopathologic examination. In the next step HybridAPC to the gastric mucosa of the fundus is applied.

SUMMARY:
Ablation of the gastric fundus mucosa with hybrid argon plasma coagulation (HYBRIDAPC) in obese patients undergoing ESG could result in restoration of ghrelin cell function in the gastric fundus. This could improve long-term outcomes in terms of body weight loss and comorbidity reduction in obese patients undergoing ESG.

DETAILED DESCRIPTION:
Obesity is one of the most prevalent diseases worldwide with a major impact on the health care system in many countries. Bariatric surgery is currently the first treatment option in obese patients because it offers lasting results on body weight loss and reduces disease-related comorbidities. In recent years, however, endoscopic sleeve gastroplasty (ESG) has emerged as a safe and effective method in treating obese patients. Considering the lower complication rate compared with bariatric surgery and the greater weight loss compared with medical therapy, ESG finds indication as a treatment in cases of class I and II obesity. In cases of BMI > 40 or higher, bariatric surgery is actually the best option to achieve lasting weight loss but may be burdened by significant morbidity and mortality related to the surgery itself. Ghrelin is a potent oressigenic hormone produced and secreted mainly by the endocrine cells of the gastric glands at the bottom of the stomach and acts in the brain to regulate food intake. Gastric ghrelin plays a key role in glucose metabolism. Obese patients generally show reduced levels of ghrelin and a high percentage of these patients are insulin-resistant, have high circulating levels of insulin, hyperglycemia or diabetes. Through gene expression data and electron microscopy the activity of GPCs (ghrelin-like cells) could be increased in obese patients and correlates with glycemic levels. A positive correlation has been suggested between ghrelin gene expression, glycemic values and body mass index in obese patients. Taken together, these data indicate that ghrelin overproduction by the stomach may be involved in the weight gain and pathogenesis of type 2 diabetes in obese patients. This study aims to demonstrate how further ablation of the gastric fundus mucosa with hybrid argon plasma coagulation (HYBRIDAPC) in obese patients undergoing ESG could result in restoration of ghrelin cell function in the gastric fundus. Indeed, HybridAPC could stimulate fundus stem cells to produce new ghrelin-secreting endocrine cells with normal secretory activity as in lean subjects. Thus normalizing ghrelin signaling to appetite/hunger areas in the brain relayed through the gut brain axis. This could improve long-term outcomes in terms of body weight loss and comorbidity reduction in obese patients undergoing ESG.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or females patients in the range of class Class I to Class II obesity (30 ≤ BMI ≤ 39.9).
* Age between 18 and 65 years (both inclusive).
* Treatment naïve for bariatric surgery or endoscopic bariatric therapy.
* Patients that have been evaluated by the local MDT and have indication to ESG.
* Willingness to comply with the substantial behavioral modifications program as required by the procedure.
* Agree to avoid any use of weight loss medications such as Meridia, Saxenda, Januvia, Xenical, or over the counter weight loss medications or supplements throughout the study.
* Women of childbearing potential should have negative urine beta human chorionic gonadotropin (hCG) pregnancy test and must agree to use acceptable contraception methods throughout the study duration.
* Able to comply with study requirements and understand and sign the Informed Consent Form.

Exclusion Criteria:

* Previous upper GI surgery (except uncomplicated cholecystectomy or appendectomy), or other endoscopic bariatric procedures or conditions,
* Prior intra-gastric balloon or another gastric implant.
* History of a structural or functional disorder of the esophagus or pharynx that may impede passage of the device such as achalasia, stricture/stenosis, esophageal varices, esophageal diverticula, esophageal perforation, severe or intractable gastro-esophageal reflux symptoms while on maximal medical therapy, uncontrolled GERD defined as LA grade C esophagitis or greater.
* History of a structural or functional disorder of the stomach including gastric polyps > 1 cm in size, gastroparesis, gastric ulcer, gastric cancer, chronic gastritis, gastric varices, hiatal hernia (>4 cm) of axial displacement of the z-line above the diaphragm.
* Active H. pylori infection (subjects with active H. pylori may continue with the screening process if they are treated with an appropriate antibiotic regimen, and eradication has been confirmed).
* Patients with history of intestinal stricture/stenosis, small bowel or colonic obstruction or any other obstructive disorder of the GI tract such as adhesive peritonitis and/or abdominal adhesions.
* Patients with any inflammatory disease (IBD).
* Autoimmune disease, including but not limited to celiac disease, or pre-existing symptoms of systemic lupus erythematosus, scleroderma or other autoimmune connective tissue disorder.
* Active hepatitis, active liver disease, hepatic insufficiency , or cirrhosis.
* Untreated/inadequately treated hypothyroidism, defined as an elevated Thyroid-Stimulating Hormone (TSH) level at Screening; if on thyroid hormone replacement therapy, must be on stable dose for at least 6 weeks prior to Screening.
* Patients with PCOS (hormonal dis-balances).
* Persistent Anemia, defined as Hemoglobin <10 g/dL.
* Significant cardiovascular disease including known history of valvular disease, or myocardial infarction, heart failure, transient ischemic attack or stroke within the last 6 months.
* Moderate or severe chronic kidney disease (CKD), with estimated glomerular filtration rate (eGFR) <45 ml/min/1.73m2 (estimated by MDRD).
* Known immunocompromised status, including but not limited to individuals who have undergone organ transplantation, chemotherapy or radiotherapy within the past 12 months, who have clinically-significant leukopenia, who are positive for the human immunodeficiency virus (HIV) or whose immune status makes the subject a poor candidate for clinical trial participation in the opinion of the Investigator.
* HbA1c > 8.5 %.
* Patients requiring exogenous insulin.
* Use of glucose-lowering drugs for diabetes mellitus treatment with the exception of sulfonylurea (SU), biguanides and sodium dependent glucose co-transporter 2 (SGLT-2) inhibitors.
* Coagulopathy, congenital or acquired intestinal telangiectasia.
* Use of systemic glucocorticoids (excluding topical or ophthalmic application or inhaled forms) for more than 10 consecutive days within 90 days prior to the Screening Visit.
* Pregnant or breast-feeding woman.
* Patients with history or current abuse of drugs or alcohol.
* Patients who are taking medications that cause weight loss such as Meridia, Saxenda, Januvia, Xenical, or over the counter weight loss medications or supplements throughout the study.
* Patients who are taking medication that cause weight gain such as anti-depressants
* Psychiatric or cooperative problems or low compliance that is a contraindication from participating in the study.
* Any health issue that might put the patient at risk if the treatment is performed, judged by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-08 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | 18 months
  Safety, Tolerability and Efficacy of HybridAPC for gastric mucosa ablation of the fundus in patients undergoing endoscopic sleeve gastroplasty
HybridAPC | 18 months
  To assess the additional effect of gastric mucosa ablation in the fundus by HybridAPC upon ESG on total body weight (Kilograms) over time

SECONDARY OUTCOMES:
Gastric Hormones | 18 months
  assess changes in plasma levels of gastric hormones. Fasting blood samples will be taken at baseline and 1, 6 and 12 months follow up visits and stored at -80℃ until assayed. Hormone measurement will be conducted using enzyme-linked immunosorbent assay (ELISA). Assay validation is performed by the manufacturer, testing the precision of the assay and its sensitivity.
  Ghrelin levels will be measured by ELISA (Lifespan Biosciences, Seattle, WA) with a sensitivity < 0.094 ng/ml and an intra- and inter-assay precision <10% and <10%, respectively.
  Leptin levels will be measured by ELISA (Lifespan Biosciences, Seattle, WA) with a sensitivity < 10 pg/ml and an intra- and inter-assay precision <6.4% and <7.4%, respectively.
  GLP-1 levels will be measured by ELISA (Lifespan Biosciences, Seattle, WA) with a sensitivity < 0.31 ng/ml and an intra- and inter-assay precision <9.09% and <8.33%, respectively.
Life changes | 18 months
  assess quality of life changes at baseline and 1,6,12 months follow up using the BAROS, SF-36 and IWQOL-Lite-CT questionnaire.
Comorbidity | 18 months
  Comorbidity improvements after ESG and Hybrid APC: Hypertension improvement was considered upon reaching values of PA < 130/80 mmHg or if antihypertensive therapy was discontinued while maintaining pressure values <130/80 mmHg. Hyperinsulinemia improvement was considered if the achieved HOMA score was < 1.8 at any time during follow-up after ESG. Type 2 diabetes mellitus (DMT2) improvement will be considered if the achieved fasting blood glucose will be on values < 126 mg/dl in at least 2 different measurements or if the glycated hemoglobin value will be < 6 % or if medical therapy will discontinue. Obstructive sleep apnea syndrome (OSAS) improvement will be considered if nocturnal pO2 > 92% or if symptoms will disappear without the use of CPAP.

CONTACTS AND LOCATIONS:
Overall Officials: ivo boskoski, Principal Investigator — Fondazione Policlinico Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Italy